CLINICAL TRIAL: NCT01580475
Title: Training, Detraining and Retraining Effects on Glycemic Control and Physical Fitness in Patients With Type 2 Diabetes
Brief Title: Training, Detraining, Retraining and Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Savvas P. Tokmakidis, Ph.D., Professor, Democritus University of Thrace
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EPEAEK - PYTHAGORAS II; 1328-5 PYTHAGORAS II (Other Grant/Funding Number: PYTHAGORAS II; co-financed by Hellenic (25%) and EC (75%))
Record Dates: First submitted 2012-03-18; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes
Keywords: glycemic control,; exercise training,; detraining,; retraining,; body composition,; strength and fitness
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle (exercise training) (Experimental): Training, detraining and retraining
  Interventions: Other: Training - detraining - retraining

INTERVENTIONS:
Other: Training - detraining - retraining — Thirteen women with type 2 diabetes followed a supervised aerobic and strength training program for 9 months, interrupted for 3 months (detraining) and resumed again for a period of 9 months (retraining).

SUMMARY:
* This study examine the effects of training, detraining and retraining, using a combined strength and aerobic exercise program, on physiological parameters in patients with type 2 diabetes.
* Thirteen women with type 2 diabetes followed a supervised aerobic and strength training program for 9 months, interrupted for 3 months (detraining) and resumed again for a period of 9 months (retraining).
* Training improved body mass index, fasting plasma glucose,postprandial glucose, glycosylated hemoglobin, peak oxygen consumption,power output and total muscle strength. Detraining reversed PPG, HbA1C and physical fitness parameters. Resumption of training however, improved further the initial training adaptations.
* Diabetic patients should follow a regular and uninterrupted exercise program throughout life in order to control glucose metabolism and improve health status.

DETAILED DESCRIPTION:
During the last decades, the positive effects of aerobic exercise in patients with type 2 diabetes have been well documented. Recently, resistance exercise has gained popularity in diabetic patients since several studies have indicated that this type of training is safe and induces favorable adaptations in physical fitness and metabolic profile. According to recent scientific evidence, a complete rehabilitation program for patients with type 2 diabetes should combine both strength and aerobic exercise; thus the American Diabetic Association in their latest guidelines recommends strength training as part of an exercise program at least two times a week.

On the contrary to the well documented effects of physical training, there is lack of data on the negative alterations of detraining in patients with type 2 diabetes. The partial or complete loss of training-induced adaptations as a consequence of training reduction or cessation is well-documented by several detraining studies in healthy subjects, older individuals and patients with coronary artery disease.

For example, the investigators know that even 6 days of physical inactivity reduces insulin action in well-trained runners which is attributed to the significant reduction in the muscle GLUT-4 level. Factors such as illness, injury, travel or vacation may interrupt the training process for longer periods, affecting the treatment in people with type 2 diabetes. For this population, it is important to quantify changes in physiological and metabolic parameters resulting from the cessation of exercise, since exercise training is a major therapeutic method.

To the best of our knowledge, there is no data concerning the loss of physiological adaptations which occurs after exercise cessation in patients with type 2 diabetes, which have previously trained for a long period of time. The current study evaluated the effects of three months of detraining after nine months of a combined strength and aerobic training program on glycemic control, body composition, peak oxygen consumption (VO2peak) and muscular strength in patients with type 2 diabetes. Further, the investigators examined the extent of the regained adaptations after the resumption of training for a period of nine months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* without micro- and macroangiopathy

Exclusion Criteria:

* type 1 diabetes
* cardiovascular disease,
* confirmed retinopathy/nephropathy/neuropathy,
* uncontrolled diabetes mellitus (HbA1c>10%).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in glycemic control measurements (follow-up for 21 months) at training (9 months), detraining (3 months) and retraining (9 months) | Changes from baseline in HbA1C, FPG and PPG at training (9 months), detraining (11 months) and retraining (21 months)
  Glycemic control was evaluated by the measurement of fasting plasma glucose (FPG), postprandial glucose (PPG) and glycosylated hemoglobin (HbA1C). PPG was calculated by the mean of four values measured at the first week of every period (baseline, 9th, 12th and 21st months).

SECONDARY OUTCOMES:
Evaluation of body composition | Changes from baseline in body composition assessment at training (9 months), detraining (3 months), retraining (9 months)
  Anthropometric Assessment: Body weight, height, BMI and waist circumference (WC).
Peak oxygen consumption (VO2peak) | Changes from baseline in VO2peak at training (9 months), detraining (11 months) and retraining (21 months)
  Measurement of Peak Oxygen Uptake: Patients underwent a symptom-limited graded exercise test on a cycle-ergometer (60 rpm). The initial load was set at 25W and increased gradually by 25W every 2-min until the patients were unable to continue. VO2peak was determined by open-circuit spirometry (E. Jaeger, IEC 601-1, Germany).
Measurement of muscular strength in patients with type 2 diabetes | Changes from baseline in muscular strength at training (9 months), detraining (11 months) and retraining (21 months)
  Muscle Strength: Maximum strength was measured with the one-repetition maximum (1 RM) method and total muscle strength was calculated as the sum of leg extension and bench press.

CONTACTS AND LOCATIONS:
Overall Officials: Savvas P. Tokmakidis, PhD, Principal Investigator — Democritus University of Thrace
Locations (1):
- Savvas P. Tokmakidis, Komotini, Greece

REFERENCES:
- [Background] Tokmakidis SP, Zois CE, Volaklis KA, Kotsa K, Touvra AM. The effects of a combined strength and aerobic exercise program on glucose control and insulin action in women with type 2 diabetes. Eur J Appl Physiol. 2004 Aug;92(4-5):437-42. doi: 10.1007/s00421-004-1174-6. PMID 15232701
- [Background] Tokmakidis SP, Volaklis KA. Training and detraining effects of a combined-strength and aerobic exercise program on blood lipids in patients with coronary artery disease. J Cardiopulm Rehabil. 2003 May-Jun;23(3):193-200. doi: 10.1097/00008483-200305000-00006. PMID 12782903
- [Background] Tokmakidis SP, Spassis AT, Volaklis KA. Training, detraining and retraining effects after a water-based exercise program in patients with coronary artery disease. Cardiology. 2008;111(4):257-64. doi: 10.1159/000127737. Epub 2008 Apr 23. PMID 18434735
- [Background] American College of Sports Medicine; American Dietetic Association; Dietitians of Canada. Joint Position Statement: nutrition and athletic performance. American College of Sports Medicine, American Dietetic Association, and Dietitians of Canada. Med Sci Sports Exerc. 2000 Dec;32(12):2130-45. doi: 10.1097/00005768-200012000-00025. PMID 11128862
- [Background] Castaneda C, Layne JE, Munoz-Orians L, Gordon PL, Walsmith J, Foldvari M, Roubenoff R, Tucker KL, Nelson ME. A randomized controlled trial of resistance exercise training to improve glycemic control in older adults with type 2 diabetes. Diabetes Care. 2002 Dec;25(12):2335-41. doi: 10.2337/diacare.25.12.2335. PMID 12453982
- [Background] Dunstan DW, Daly RM, Owen N, Jolley D, De Courten M, Shaw J, Zimmet P. High-intensity resistance training improves glycemic control in older patients with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1729-36. doi: 10.2337/diacare.25.10.1729. PMID 12351469